CLINICAL TRIAL: NCT06097689
Title: A Pilot Study to Assess the Feasibility of a Novel Non-Invasive Technology to Measure Glucose Dynamics in Adults Living with Type 1 Diabetes Mellitus: a Single-Arm Pilot Study
Brief Title: A Pilot Study to Assess the Feasibility of a Novel Non-invasive Technology to Measure Changing Blood Glucose Levels in Adults with Type-1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liom Health AG (Industry)
Collaborators: DCB Research AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SPN-005
Record Dates: First submitted 2023-10-10; First posted 2023-10-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes Mellitus; Type 1 Diabetes Mellitus with Hypoglycemia; Type 1 Diabetes Mellitus with Hyperglycemia
Keywords: Hypoglycemia; Hyperglycemia; Diabetes; Transcutaneous; Spectral fingerprint; Noninvasive
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational arm (Experimental): Induction of different glycaemia states via intravenous regular insulin and intravenous glucose administration and measurements of transcutaneous spectral data with the investigational device and reference blood glucose values.
  Interventions: Device: Lab Demo 1.0

INTERVENTIONS:
Device: Lab Demo 1.0 — Lowering of the participants blood glucose with the application of insulin to induce hypoglycaemia, followed by the application of glucose to induce hyperglycaemia and finally insulin to restore euglycemia.
  During the different glycaemia states, transcutaneous spectral data are collected continuously with the device and paired with reference measurements (venous blood and interstitial fluid).

SUMMARY:
The primary aim of this study is to assess the feasibility of the Lab demo 1.0 and associated computational models to detect and track glucose changes noninvasively and transcutaneously in defined and dynamic states of glycemia.

ELIGIBILITY:
Inclusion Criteria:

* 1.1nformed Consent signed by the subject
* 1.2 Male and female subjects 18 - 60 years of age (inclusive)
* 1.3 Skin colour Type I, II, or III according to Fitzpatrick Scale (see Appendix 1)
* 1.4 Type 1 diabetes diagnosed > 12 months ago
* 1.5 Intensified insulin therapy scheme using multiple daily injection (MDI) or continuous subcutaneous insulin infusion (CSII) for more than 6 months
* 1.6 BMI between 18.5 and 28.0 kg/m2
* 1.7 Using a CGM/FGM system (Freestyle Libre2, Freestyle Libre3, Dexcom G6 or Dexcom G7)
* 1.8 Willingness to follow the study procedure

Exclusion Criteria:

* 2.1 In female subjects: pregnancy or breastfeeding period (self-reported)
* 2.2 HbA1c of > 9.0% (based on last measurement by treating physician but not older than 120 days) Note: To be repeated at the study site if measurement is older than 120 days or not available
* 2.3 History of cardiovascular diseases
* 2.4 Irregular 12-lead ECG upon investigator's judgement
* 2.5 Medical history of epilepsy or other neurological disease associated with seizure events
* 2.6 Atypical skin condition (e.g., Hyperkeratosis, Hyperpigmentation) or presence of tattoos or scars in the measurement area (wrist) that could impair validity of measurement upon investigator's judgement
* 2.7 Known sensitivity to medical grade adhesives or other skin-related complications, which might influence the outcome
* 2.8 Not able to understand, write or read German
* 2.9 Participation in another investigation with an investigational drug within the 30 days preceding and during the present investigation
* 2.10 Enrolment of the PI, his/her family members, employees and other dependent persons

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Changes in spectral fingerprints measured by the Lab Demo 1.0 at fluctuations of venous blood glucose levels | The data is collected during the study procedure (6 to 8 hours)
  The primary outcome is to assess the feasibility/capacity of the prototype device to measure changes in spectral fingerprints at fluctuations of venous blood glucose levels in ranges of hypoglycaemic and hyperglycaemic states.

SECONDARY OUTCOMES:
Changes in spectral fingerprints measured by the Lab Demo 1.0 at fluctuations of interstitial fluid glucose levels | The data is collected during the study procedure (6 to 8 hours)
  The secondary outcome is to assess the feasibility/capacity of the prototype device to measure changes in spectral fingerprints at fluctuations of interstitial fluid glucose levels in ranges of hypoglycaemic and hyperglycaemic states.
Spectral fingerprints measured by the Lab Demo 1.0 | The data is collected during the study procedure (6 to 8 hours)
  This secondary objective consists of describing the spectral fingerprints at different blood glucose levels (defined by both venous blood glucose and interstitial fluid glucose)
Blood glucose levels | During the study procedure (6 to 8 hours)
  Blood glucose levels at the time of changes in spectral fingerprints measured by the Lab Demo 1.0
Heart rate | During the study procedure (6 to 8 hours)
  Heart rate at the time of changes in spectral fingerprints measured by the Lab Demo 1.0
Oxygen saturation | During the study procedure (6 to 8 hours)
  Oxygen saturation at the time of changes in spectral fingerprints measured by the Lab Demo 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Rebeaud, PhD, Study Director — Liom Health AG; Markus Laimer, Prof Dr med, Principal Investigator — University Department of Diabetology, Endocrinology, Nutritional Medicine & Metabolism (UDEM), Inselspital, Bern University Hospital
Locations (1):
- Markus Laimer, Bern, Canton of Bern, Switzerland